CLINICAL TRIAL: NCT03625739
Title: Population Pharmacokinetics of Anti-tuberculosis Drugs in Children With Tuberculosis
Status: Recruiting | Type: Observational
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Shandong University (Other); Hopital Universitaire Robert-Debre (Other); Rennes University Hospital (Other)
Responsible Party: Principal Investigator, Adong Shen, Deputy Chief of China National Clinical Research Center for Respiratory Diseases, Beijing Children's Hospital
Other Study IDs: BCH_PPK003
Record Dates: First submitted 2018-08-08; First posted 2018-08-10 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Antitubercular Agents; Isoniazid; Rifampin; Pyrazinamide; Ethambutol; Levofloxacin; Moxifloxacin; Gatifloxacin; Amikacin; Capreomycin; Kanamycin; Streptomycin; Ethionamide; Cycloserine; terizidone; Clofazimine; bedaquiline; OPC-67683; Aminosalicylic Acid; Amoxicillin-Potassium Clavulanate Combination; Thioacetazone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Biospecimen Retention: Samples With DNA — whole blood and plasma
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: anti-tuberculosis drug — The intervention drugs are prescribed by treating caregiver
  Other Names: Isoniazid; Rifampicin; Pyrazinamide; Ethambutol; Levofloxacin; Moxifloxacin; Gatifloxacin; Amikacin; Capreomycin; Kanamycin (Streptomycin); Ethionamide; Cycloserine; terizidone; Clofazimine; Bedaquiline; Delamanid; p-aminosalicylic acid; Imipenem-cilastatind; Amoxicillin-clavulanate; Thioacetazone

SUMMARY:
This study is based on the hypothesis that the pharmacokinetics of anti-tuberculosis drugs in TB children are different from adults. The investigators aim to study the population pharmacokinetics of children receiving the anti-tuberculsis drugs for treatment of TB. In this study, the investigators will detect drug concentration in plasma by using residual blood samples of blood gas analysis and other clinical tests and employ computers for constructing population pharmacokinetic models. In addition, the investigators also want to correlate use of anti-tuberculsis drugs with treatment effectiveness and incidence of adverse effects in children. This novel knowledge will allow better and more rational approaches to the treatment of TB in children. It will also set the foundation for further studies to improve anti-tuberculosis drug therapies for children.

DETAILED DESCRIPTION:
1.Establish population pharmacokinetic (PPK) models of each anti-tuberculsis drug in children by nonlinear mixed effect modeling (NONMEM).

1. At different timepoint after anti-tuberculsis drug administration, plasma samples of 100 children will be collected from neonatal intensive care unit (NICU) and pneumology department for each drug. The clinical information includes demography, medication, concentration data, blood biochemical parameters and so on .
2. Plasma samples will be tested by high performance liquid chromatography (HPLC).
3. PPK models of anti-tuberculsis drug will be established by NONMEM program.
4. The reliability and stability of the PPK model will be evaluated by 1000 times of Bootstrap procedure and normalized predictive distribution error (NPDE).

2.Evaluation of the clinical feasibility and safety of individualized dosing.

1. According the results of PPK models, the investigators will use dosages recommended in models to cure TB children in prospective studies. For anti-tuberculsis drug, 50 children will be collected.
2. The investigators will compare the therapeutic effects and safety between children with conventional therapies and children with individualized therapies, including proportions of children with effective drug concentration, improvement speed of of children, liver and kidney functions of of children, adverse reactions of drugs and so on.

ELIGIBILITY:
Inclusion Criteria:

* Children (0-18 years old) with anti-tuberculosis therapy against TB.
* The anti-tuberculsis therapy includes drugs commonly used in children infectious diseases
* Informed consent signed by the parents and/or guardians.

Exclusion Criteria:

* Anti-tuberculosis drugs aren't involved in the therapies of children.
* It is unable to provide complete medical records or the current condition cannot accept the study process.
* Patients are allergic to anti-tuberculsis drugs.
* Parents and/or guardians do not agree to participate in this study.

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with anti-tuberculosis therapies.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
maximum concentration (Cmax) | up to 4 weeks
  Cmax is a term used in pharmacokinetics refers to the maximum (or peak) serum

SECONDARY OUTCOMES:
time to achieve maximum concentration (Tmax) | up to 4 weeks
  Tmax is the term used in pharmacokinetics to describe the time at which the Cmax
absorption rate constant (ka) | up to 4 weeks
  Ka is the rate constant of drug absorption.
elimination rate constant (kel) | up to 4 weeks
  The elimination rate constant is a value used in pharmacokinetics to describe the rate at which a drug is removed from the system.
half-life (t1/2) | up to 4 weeks
  Half-life is the time required for a quantity to reduce to half its initial value.

CONTACTS AND LOCATIONS:
Overall Officials: A-Dong Shen, Master, Principal Investigator — Beijing Children's Hospital of Capital Medical University; Yu-Jie Qi, Master, Study Director — Beijing Children's Hospital of Capital Medical University; Wei Zhao, Doctor, Study Director — Children's Hospital of Hebei Province;Shandong Provincial Qianfoshan Hospital
Locations (1):
- Beijing Children's Hospital of Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Jacqz-Aigrain E, Leroux S, Zhao W, van den Anker JN, Sharland M. How to use vancomycin optimally in neonates: remaining questions. Expert Rev Clin Pharmacol. 2015;8(5):635-48. doi: 10.1586/17512433.2015.1060124. Epub 2015 Aug 4. PMID 26289222
- [Background] Ho PL, Lo PY, Chow KH, Lau EH, Lai EL, Cheng VC, Kao RY. Vancomycin MIC creep in MRSA isolates from 1997 to 2008 in a healthcare region in Hong Kong. J Infect. 2010 Feb;60(2):140-5. doi: 10.1016/j.jinf.2009.11.011. Epub 2009 Dec 2. PMID 19961873
- [Background] Kearns GL, Abdel-Rahman SM, Alander SW, Blowey DL, Leeder JS, Kauffman RE. Developmental pharmacology--drug disposition, action, and therapy in infants and children. N Engl J Med. 2003 Sep 18;349(12):1157-67. doi: 10.1056/NEJMra035092. No abstract available. PMID 13679531